CLINICAL TRIAL: NCT02041611
Title: Prospective Evaluation of T-cell Immune Status in Patients With Newly Diagnosed High Grade Gliomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: J1389; NA_00086826 (Other: JHMIRB)
Record Dates: First submitted 2014-01-10; First posted 2014-01-22 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: High Grade Glioma
Keywords: WHO grade III and IV
MeSH Terms: conditions — Glioma; Lymphoma, Follicular | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Standard Care Pts Eval of T-Cell Immune Status (Other): Pts undergoing standard radiation/TMZ and adjuvant TMZ will have blood collections at 6 different time points throughtout their treatment to evaluate T Cell changes
  Interventions: Procedure: Blood collections

INTERVENTIONS:
Procedure: Blood collections — pts will have 6 blood collections (30ml/collection) throughout course of standard treatment

SUMMARY:
The primary goal of this study is evaluate T cell immune status and immune reconstitution and the association with specific cytokines in patients with newly diagnosed HGGs undergoing the standard RT/TMZ and adjuvant TMZ.

DETAILED DESCRIPTION:
Numbers of T-cell subtypes at six time points in patients with newly diagnosed HGGs undergoing standard RT/TMZ and adjuvant TMZ:

1. Baseline within 2 weeks before initiation of RT/TMZ
2. At the end of RT/TMZ approximately week 6
3. Before adjuvant TMZ approximately week 10
4. After 2 cycle of TMZ approximately week 18
5. After 4 cycle of TMZ approximately week 26
6. Three month after last cycle of TMZ

Secondary Endpoints

1. Changes in serial T cell subtypes and cytokines levels
2. Incidence of lymphopenia related infections
3. Changes in T-cell numbers and subtypes with TMZ administration
4. Overall survival

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be at least 18 years of age.
2. Patients must have histologically confirmed new diagnosed high grade glioma by pathology (WHO grade III and IV).
3. Patients proposed post-operative treatment plan must include standard radiation and temozolomide.
4. Patients must have a Karnofsky performance status ≥ 60% (i.e. the patient must be able to care for himself/herself with occasional help from others).
5. Patients must be able to provide written informed consent.
6. Steroid use is allowed.

Exclusion Criteria:

1. Patients with HIV are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-07-13 (Actual); Primary Completion 2013-09-02 (Actual); Study Completion 2015-12-17 (Actual)

PRIMARY OUTCOMES:
Changes in T Cell subtypes and cytokines as a function of treatment | 6 time points in pts undergoing standard RT/TMZ and adjuvant TMZ
  baseline approx 6wks approx 10wks aprox 18wks approx 26wks 3 months after last cycle of TMZ

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A Grossman, MD, Study Chair — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins, Baltimore, Maryland
  - Washington University, St Louis, Missouri